CLINICAL TRIAL: NCT05258344
Title: Evaluation of the Reliability and Validity of The '6 Minute Pegboard and Ring Test' Unsupported Arm Function Exercise Test in Patients With Breast Cancer
Brief Title: Reliability and Validity of The '6 Minute Pegboard and Ring Test' in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO 22/41
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Functional Performance; Upper Extremity
Keywords: breast cancer; 6 Minute Pegboard and Ring Test; Arm exercise endurance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is one of the most common cancers among women in the world and its incidence reaches up to 16%.Although survival can be increased with early diagnosis and more effective therapies, physical complications such as lymphedema, upper extremity dysfunction and chronic pain are frequently seen during and/or after breast cancer treatments. It has been determined that lymphedema associated with breast cancer treatment is a factor that mediates and/or exacerbates the adverse effects of breast cancer treatments on upper extremity functional capacity and quality of life of patients.It was determined that the 6 Minute Pegboard and Ring Test (6PRT) score showed a clear relationship with the upper extremity daily living activities (ADLs), and it was concluded that the 6 Minute Pegboard and Ring Test (6PRT) test could be used as an appropriate test in pulmonary rehabilitation programs to predict and show the improvement of daily living activities (ADLs). Therefore, in this study; The results to be obtained by evaluating the validity and reliability of the 6 Minute Pegboard and Ring Test (6PRT) test in breast cancer patients will increase the use of this test in both testing arm endurance and arm exercise capacity in breast cancer patients, and predicting the effect on daily living activities (ADLs)

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers in the world and it can be diagnosed as high as 16 percent. According to a 2016 report published by the Ministry of Health, the incidence of breast cancer in Turkey is 46.8 per 100,000 people and 17,000 women are diagnosed with breast cancer each year. While breast cancer survival rate is 80 percent in developed countries, it varies between 40 and 60 percent in low-middle income countries. While early diagnosis and more effective therapies may improve survival time, physical complications such as lymphedema, upper extremity dysfunctions and chronic pain are frequent during and/or following breast cancer treatments. Breast cancer treatment-related lymphoma is one of the most common complications that scare and disturb patients. In the report of the International Society of Lymphology (ISL), lymphedema is defined as a disease that occurs as a result of water, plasma proteins, extravascular fluid and parenchymal cell accumulation in the interstitial area depending on the low transport capacity of the lymphatic system. In secondary lymphedema, the reduced carrying capacity is usually associated with surgical, chemotherapy and/or radiotherapy related cancer treatments. The incidence of secondary upper limb lymphedema related to breast cancer treatment was found to be 16%. In the latest clinical guide on the assessment and treatment of lymphedema after the treatment of breast cancer, the risk factors of lymphedema are examined in three groups: treatment-related, patient-related and disease-related risk factors. Risk factors associated with the treatment; axillary lymph node dissection, mastectomy, excessive removal of lymph nodes, radiotherapy and chemotherapy. Patient-related risk factors include body mass index values of 30 or above, lack of regular physical activity and exercise, and changes in weight gain after surgery. Finally, the risk factor related to the disease has been reported as the presence of metastatic lymph nodes. After the breast cancer treatment, although a good level of functional improvement is observed in most patients, it is stated that the effects of these treatments on functional capacity, daily life, work and social activities and quality of life may be significant and long-lasting. Further, it has been established that lymphedema related to breast cancer treatment is a factor that mediates and/or exacerbates the negative effects of breast cancer treatments on functional capacity and on the quality of life of patients. Furthermore, as the intensity of lymphoma increases in patients with lymphedema related to breast cancer treatment, there is also an increase in emotional state changes such as stress, anxiety and fear. Upper extremity lymphedema, developed following breast cancer treatment, usually affects glenohumeral joint by increasing the stress in the tendons of the rotator cuff muscles and disrupting the scapulohumeral rhythm. Additionally, lymphedema may cause symptoms such as a decrease in muscle strength and mobility width of upper extremity, pain and fatigue and as a result may result in reduction of activity limits and functional level of upper extremity. Another factor in reducing the capacity of the upper extremity is the development of kinesiophobia related to the affected extremity in patients. Patients are able to restrict the use of extremity to prevent exacerbation of lymphedema. The reduction in functional capacity following breast cancer treatment is frequent but as far as we know there is no validated functional test to assess upper limb exercise capacity. Given that the number of women living with breast cancer increases every year, the existence of an objective clinical test for upper limb function may be a useful evaluation method.

"6 Minute Pegboard and Ring Test (6PRT)" is a valid and reliable, practical and easy-to-use test that assesses unsupported arm endurance in patients with chronic obstructive pulmonary disease (COPD), asthmatic patients and healthy persons. For the test, patients are asked to carry as many rings as possible within 6 minutes and the number of rings carried over for 6 minutes is recorded as a score. A study in patients with mild-to-very severe chronic obstructive pulmonary disease (COPD) has shown a positive association between the 6PRT score and the activity counts assessed by an accelerometer. Furthermore, it has been established that the 6PRT score represents a clear association with the upper extremity daily living activities (ADLs) and it has been concluded that the 6PRT test can be used as an appropriate test for the prediction and development of daily living activities (ADLs) in pulmonary rehabilitation programs. As a result, in this study; Results based on assessing the validity and reliability of the 6PRT test for breast cancer patients will increase the use of the test to predict the effect on daily living activities (ADLs) in patients with breast cancer, both on arm endurance and arm exercise capacity.

Demographic information: name, age, diagnosis, medical history (months of surgery), release form of lymphoma, treatments for lymphoma, radiotherapy (number of days), chemotherapy (number of cycles), surgical type (lumpectomy, segmental mastectomy, modified radical mastectomy, radical mastectomy), body weight, height, BMI dominant and affected side, curriculum vitae (CV), family history, lifestyle traits (smoking, exercise habit) will be recorded.

Arm length, arm and underarm circumference: We analyzed that your participants perimeter and length measurements of dominant side arms shall be measured using a measuring tape. If participants have developed lymphedema, the extremities of the related party will not be evaluated. Length of the arm shall be measured from acromion- to lateral limit of radial styloid process when the arm is in anatomic position. The radius of the arm shall be measured from the mid-zone between the acromion and the olecranon, around the forearm as well as the area where the arm reaches its largest diameter while it is relaxed near the body.

Evaluation of the Hand Grip Force: The hand gripping force shall be measured with the person bent by an elbow in a sitting position with his/her back vertically upright (the person's arm is attached to the body, in a neutral position and the elbow bent by 90 degrees, the wrist is neutral). For the dominant and non-dominant side measurements shall be repeated three times. Three measurements shall be averaged for both sides and recorded in Newtons (N).

Assessment of Shoulder Joint Movement Openness: Shoulder, flexion, extension, abduction, internal and external rotation joint mobility openings shall be measured actively and/or passively and the results shall be recorded as "limited" or "no limitations."

Pain Threshold Assessment: The pain threshold evaluation is performed by an algometer ('J tech Algometer', USA), from the region located in the volar region of the forearm, 10 cm distal of the medial and lateral epicondylar middle point in both upper limbs. With the 1 cm2 head of the algometer, vertical pressure will be applied to the application area and the patient will be asked to say "Yes" when they feel pain with the pressure applied. The measurement will be repeated 3 times and the pressure pain threshold values will be recorded taking the arithmetic mean of the three trials. Algometer measurement of pain threshold is a non-invasive and reliable method used in literature.

Information related to lymphedema: Individuals' lymphoma effects ("present", "none") will be questioned and recorded. Lymphedema duration will be recorded numerically (years).

Evaluation of Lymphedema: The environmental measurement shall be performed separately at both upper extremities, with a mild pressure at the patient sitting, with the forearm supination, elbow full extension and arm at 90 degrees abduction, with a non-stretching measuring tape. Peripheral measurement will be performed at ulnar styloid level in the wrist and at five cm intervals from this level to axilla. According to the environmental measurement, women with a minimum difference of 2 cm between the affected and the unaffected side are considered positive for lymphedema. The affected and unaffected arm volumes shall be calculated using the cut comfort formula (frustum method). Considering the difference between dominant and non-dominant arm volumes, 3.3% volume correction will be applied in women that have a dominant arm effect. The severity of lymphedema will be determined according to the differences between the affected and unaffected arms on volumetric measurements (calculated using frustum method). (mildly severe lymphedema: 200-<250 ml difference; moderate-severe lymphedema: 250-<500 ml difference: severe lymphedema: >500 ml difference).

Evaluation of Upper Extremity Functionality: Individual upper-limb functionality will be evaluated in the "Questionnaire Disability of Arm, Shoulder and Hand (DASH)" which is a short version of the "Questionnaire Quick Disability of Arm, Shoulder and Hand (Q-DASH-T). It comprises 38 statements in total and 3 subdivisions including function/symptom, business model and musicians model. The Committee assesses problems in daily life and social life, pain, neurological symptoms and problems in work and sleep patterns. The scoring is performed using a five-stage likert scale. Scoring of the upper limb events according to this scale; 1-there is no difficulty, 2-mild difficulty, 3-moderate difficulty, 4-excessive difficulty, 5-not being able to do it at all. The total score is calculated using the formula "[(total score of items marked/number of items marked)-1]x25" and ranges from 0-100. "0" is the score in which the functions are not affected at all and "100" is where the functions are maximum.The Questionnaire Quick Disability of Arm, Shoulder and Hand (Q-DASH-T) is the short version of Questionnaire Disability of Arm, Shoulder and Hand (DASH) consisting of 11 questions. The scoring system is same as the long version.

Assessment of Unsupported Arm Exercise Capacity and Arm Function/Endurance: Will be assessed in "6 minute Pegboard and Ring Test-6PRT." During the test, the patient is asked to sit in front of a perforated panel and for 6 minutes to move as many rings as possible, using both hands simultaneously, from two bottom holes to two upper holes. The test is run with the test by putting on a few rings before the test. Standardized encouragement is provided every minute during the test. The number of rings carried over for 6 minutes constitutes the final score. Before and after the test, pulse oximeter questions heart rate and oxygen saturation, dyspnea with modified Borg scale, overall fatigue and arm fatigue detection. For the validity of the test, the test will be repeated in the same conditions as one week apart in the same patient.

Maximal Arm Exercise Capacity Assessment: An exercise test with an arm ergometer and a maximal symptom with a limited exercise test will be evaluated and the reliability of the 6PRT test will be used as criterion.

Evaluation of Upper Extremity Muscle Endurance: The first and second subtests of the Functional Impairment Test Hand, and Neck/Shoulder/Arm (FIT-HaNSA) test will be used to assess the upper limb muscle endurance of the individuals and will be used as criteria for the reliability of the 6PRT test. The test will be performed bilateral. During the test, the patient will be asked to place three 1 kg bottles at 10 cm intervals first on a 25 cm shelf at waist level and on the other shelf at 25 cm height, resting on a 60 pulse metronome per minute until they feel that they cannot continue for 5 minutes. Then they will be asked to place the bottles in the same manner on a shelf located 25 cm below a shelf at eye level. Patients' total time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-80,
2. Volunteering to participate in the research,
3. At least 15 months after breast cancer surgery,
4. 6 months after active breast cancer treatment (ie surgery/chemotherapy)
5. Having no problem in reading and/or understanding the scales and being able to cooperate with the tests.

Exclusion Criteria:

1. Presence of active infection,
2. Presence of bilateral breast cancer,
3. Presence of a history of surgical, neurological or orthopedic problems that may affect upper extremity functionality other than breast cancer surgery,
4. Having a neurological disease or other clinical diagnosis that may affect cognitive status,
5. Having musculoskeletal and neurological disease, symptomatic heart disease, previous lung surgery and malignant disease that may affect exercise performance.
6. Presence of unstable hypertension or diabetes mellitus

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-80 who were diagnosed with breast cancer in Hacettepe University Hospital, Department of Internal Medicine, Department of Medical Oncology and volunteered to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
6 minute Pegboard and Ring Test - 6PRT | one year
  Total number of rings installed within six

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided